CLINICAL TRIAL: NCT02213120
Title: To Study the Characteristics of Different Types of Vertigo in Patients Attending the ENT Clinics.
Brief Title: To Study the Characteristics of Different Types of Vertigo in Patients Attending the Ear Nose & Throat (ENT) Clinics.
Acronym: VERTIGO
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Dimension Research (Industry)
Responsible Party: Sponsor
Other Study IDs: BETA5003
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Vertigo
Keywords: Vertigo, Dizziness
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dizziness: Patients with Dizziness

SUMMARY:
The VERTIGO study is likely to help determine characteristics of different types of vertigo in patients presenting in the Ear Nose & Throat (ENT) clinics with complaints of dizziness. Moreover, it will also help to develop an understanding about the current management practices of this condition at local level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age and older
* Patients with vestibular vertigo of known or unknown origin
* Patients who are willing and able to provide written informed consent

Exclusion Criteria:

* Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion based on clinical judgment
* Patient with psychiatric disorders, significant neurological disorder or spinal cord damage that would make the evaluation difficult for the investigator
* Patients who are not willing to give informed consent
* Patients with a known history of hypersensitivity to betahistine
* Patients with a history of pheochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic/Private Clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Characteristics (Different Types) of dizziness | 6 months
  It will be determined that a patient with dizziness is suffering from what type of Vertigo i.e. Benign Paroxysmal Positional Vertigo, Menier's Disease, Vestibular Neuritis, Labyrinthitis or any other. As these are clinical types of Vertigo these cannot be measured in units

SECONDARY OUTCOMES:
Quality of Life (QoL) of patients at baselines | 6 months
  Dizziness Handicap Inventory will be used
Management of vertigo currently in practice | 6 months
  As per practice of the physician/Investigator. Management of Vertigo is either by certain maneuvers such as Epley's and Simont or by medications. For the maneuvers, no unit can be defined. The information for medication which will be collected will be Name (preferably the generic name), Dose, Units (form of the medicine), Route and Frequency.
QoL of patients post treatment | 6 months
  Dizziness Handicap Inventory will be used

CONTACTS AND LOCATIONS:
Overall Officials: Raeefuddin Ahmed, MD, Study Director — Abbott
Locations (11):
- Pakistan (11):
  - Research facility ID ORG-001139, Hyderābād
  - Research facility ID ORG-001053, Islamabad
  - Research facility ID ORG-001070, Karachi
  - Research facility ID ORG-001051, Karachi
  - Research facility ID ORG-001069, Karachi
  - Research facility ID ORG-001050, Karachi
  - Research facility ID ORG-001060, Lahore
  - Research facility ID ORG-001054, Lahore
  - Research facility ID ORG-001055, Lahore
  - Research facility ID ORG-001061, Lahore
  - Research facility ID ORG-001052, Peshawar